CLINICAL TRIAL: NCT00743561
Title: Study of the Performance of Ambulatory Nocturnal Polygraphy in the Diagnosis of Sleep Apnea in Multiple System Atrophy
Brief Title: Assessment of Ambulatory Polygraphy in the Detection of Sleep Apnea in Multiple System Atrophy (SAMSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHUBX - 2007/04
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Sleep Apnea Syndromes; Multiple System Atrophy
Keywords: MSA; sleep apnea; ambulatory polygraphy; polysomnography
MeSH Terms: conditions — Sleep Apnea Syndromes; Multiple System Atrophy | interventions — Polysomnography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Device: Polysomnography; Device: ambulatory polygraphy

INTERVENTIONS:
Device: Polysomnography — Simultaneous recording of electro-encephalography, tibial and submental electro-myography, electro-oculography, nasal air flow, oxygen saturation, as well as the thoracic and abdominal respiratory effort
Device: ambulatory polygraphy — Simultaneous recording of nasal air flow, oxygen saturation, as well as the abdominal and thoracic respiratory effort.

SUMMARY:
The purpose of this study is to determine whether ambulatory polygraphy during a short hospitalization in a neurology unit has the same performance than inpatient polysomnography, the actual gold standard, in the diagnosis of sleep apnea in patients suffering from multiple system atrophy (MSA).

DETAILED DESCRIPTION:
MSA patients frequently show sleep apnea. Inpatient polysomnography is currently the gold standard in the diagnosis of sleep apnea. However, its limited availability and high costs restrain a systematic screening of MSA patients. In contrast, ambulatory polygraphy is easy to achieve during a short hospitalization in a neurology unit or at the patient's home. Its validity in MSA is unknown.

The purpose of this study is to assess whether ambulatory polygraphy realized during a short hospitalization in a neurology unit has the same performance than inpatient polysomnography in the diagnosis of sleep apnea in MSA patients. Polygraphy recordings will also be done during daytime to characterize diurnal respiratory disturbances.

Principal Objective :

To assess the performance of ambulatory polygraphy in the diagnosis of sleep apnea in MSA patients in comparison to polysomnography (reference test).

Secondary Objectives :

To assess the performance of ambulatory polygraphy in the diagnosis of sleep apnea in comparison to polysomnography in two subgroups of MSA patients: one at high risk and one at low risk according to the results of the Berlin Questionnaire and the Epworth Sleepiness Scale.

To assess the inter-rater agreement of ambulatory polygraphy. To assess the association between sleep apnea and (i) the severity of MSA, (ii) the quality of life, (iii) the quality of sleep, and (iv) the presence of depression.

To assess the association between the severity of sleep apnea and (i) the severity of MSA, (ii) the quality of life, (iii) the quality of sleep and (iv) the presence of depression.

To assess diurnal respiratory disturbances in MSA by performing polygraphical recordings during daytime.

To assess the association of diurnal respiratory disturbances in MSA and (i) the severity of MSA and (ii) the quality of life.

Study design :

Cross-sectional prospective study (delay of one month between ambulatory polygraphy during a short hospitalization in a neurology unit and inpatient polysomnography). Each test will be carried out an interpreted blind to the other test.

Study plan:

Visit of Selection (V0)

* Verification of eligibility
* Study related information Visit of inclusion (From 0 to 90 days after selection)
* Verification of eligibility
* Diagnosis criteria
* Oral informed consent of patient or representative
* Clinical examination by using UMSARS, MMSE, Berlin Questionnaire, Epworth Sleepiness Scale, PSQI, MSA-QoL, SF-36 and Beck Depression Inventory
* Ambulatory polygraphy during a short hospitalization in a neurology unit Visit of follow-up (V2, 1 month ± 5 days after V1)
* Clinical examination by using UMSARS, Berlin Questionnaire and Epworth Sleepiness Scale
* Inpatient polysomnography

Number of subjects :

30 patients (estimation of 15 patients at high risk of having sleep apnea and 15 patients at low risk).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of "probable" MSA according to current consensus criteria (Gilman et al. 1999, PMID 10223419)
* Age 30-80 years
* Oral informed consent of patient or representative
* Patient requiring hospitalization in a neurology unit

Exclusion Criteria:

* Progressive cancer
* Significant cognitive impairment (MMSE<24)
* Sleep apnea
* Respiratory disorder
* Less than one year since previous polysomnography or ambulatory polygraphy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the performance of ambulatory polygraphy in the diagnosis of sleep apnea in comparison to polysomnography. Sensitivity, specificity, positive and negative predictive values, positive and negative likelihood ratios will be calculated. | 1 month

SECONDARY OUTCOMES:
Assessment of the performance of ambulatory polygraphy in the diagnosis of sleep apnea in comparison to polysomnography in two subgroups (high vs low risk for sleep apnea). Performances of the tests will be compared between the two sub-groups. | 1 month
Assessment of the performance of ambulatory polygraphy in the diagnosis of sleep apnea in comparison to polysomnography for different AHI thresholds (ROC curve analysis). | 1 month
Assessment of inter-rater variability by (i) calculating the intraclass correlation coefficient and its confidence interval (95%) for estimation of apnea/hypopnea index, and (ii) calculating kappa coefficient for SAOS diagnostic (dichotomous variable). | 1 month
Assessment of the association between sleep apnea and: severity of MSA (UMSARS), quality of life (MSA-Qol, SF-36), quality of sleep (PSQI) and depression (BDI). | 1 month
Assessment of the association between the severity of sleep apnea and: severity of MSA (UMSARS), quality of life (MSA-Qol, SF-36), quality of sleep (PSQI) and depression (BDI). | 1 month
Assessment of diurnal respiratory disturbances: 1. calculation of the AHI and the indices of obstructive and central respiratory events; description of all type of abnormal respiratory pattern. | 1 month
Assessment of the association between diurnal respiratory disturbances and: 1. the severity of MSA as measured by the UMSARS 2. the quality of life as measured by the MSA-QoL and SF-36 | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Wassilios Meissner, MD PhD, Principal Investigator — University Hospital Bordeaux, France; Paul PEREZ, MD, PhD, Study Chair — USMR, University Hospital, Bordeaux
Locations (2):
- France (2):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - CHU de Bordeaux - Hôpital du Haut-Lévêque - Département de Neurologie - Centre de référence nationale maladie rare AMS, Pessac